CLINICAL TRIAL: NCT06687343
Title: The Importance of Non-essential Amino Acids for Maintaining Skeletal Muscle Protein Synthesis Rates in Healthy Young Men
Acronym: NEAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL83031.068.22 / METC22-074
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy Males
Keywords: muscle protein synthesis; amino acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EAA + NEAA (Active Comparator): Dietary intake of both EAA and NEAA, representing a normal diet
  Interventions: Dietary Supplement: EAA Supplement; Dietary Supplement: NEAA Supplement
- EAA + maltodextrin (Experimental): Dietary intake of EAA, with NEAA replaced by maltodextrin
  Interventions: Dietary Supplement: EAA Supplement; Dietary Supplement: Maltodextrin Supplement
- EAA (Experimental): Dietary intake of EAA, with NEAA replaced by additional EAA
  Interventions: Dietary Supplement: EAA Supplement

INTERVENTIONS:
Dietary Supplement: EAA Supplement — Dissolved in water and ingested 4 times a day
Dietary Supplement: NEAA Supplement — Dissolved in water and ingested 4 times a day
  Arms: EAA + NEAA
Dietary Supplement: Maltodextrin Supplement — Dissolved in water and ingested 4 times a day
  Arms: EAA + maltodextrin

SUMMARY:
Background: Protein intake is important for maintaining skeletal muscle mass. These proteins consist of a collection of small building blocks which are called amino acids. There are two types of amino acids that are needed to build muscle: essential amino acids (EAA) and non-essential amino acids (NEAA). EAAs cannot be made in the body and must be consumed through foods, while NEAAs can be made within the body. However, if NEAA are not consumed through foods, the process of making NEAA in the body costs the body energy. It is still unknown what the impact of a diet containing too few non-essential amino acids is for muscle building and the body's energy metabolism.

Objective: To determine if a diet lacking NEAA, with or without being replaced by additional EAA, influences muscle protein building and whole-body metabolism.

Study design: Randomized, parallel design, double-blind, 10-day dietary intervention study.

Study population: 45 healthy (BMI 22-30 kg/m2) young males (age: 18-35 y inclusive).

Hypothesis: It is hypothesized that a diet lacking NEAA, with or without being replaced by additional EAA, decreases muscle protein building in humans.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18 and 35 y inclusive
* BMI between 22 and 30 kg/m2
* Non-smoker
* Having given informed consent

Exclusion Criteria:

* Participating in a structured (progressive) exercise program
* Smoker
* Diagnosed GI tract disorders or diseases
* Diagnosed musculoskeletal disorders
* Diagnosed metabolic disorders (e.g. diabetes)
* Cardiovascular disease
* Hypertension (blood pressure above 140/90 mmHg)
* Donated blood 3 months prior to test day
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories).
* Chronic use of gastric acid suppressing medication
* Chronic use of anti-coagulants
* Any intolerance to foods included in the standardized diet intervention
* Any implants that would be a contra-indication for performing an MRI scan

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Integrated skeletal muscle protein fractional synthesis rates | 10 days
  Calculated by the change in deuterium labelled alanine in skeletal muscle protein

SECONDARY OUTCOMES:
Integrated skin protein fractional synthesis rates | 10 days
  Calculated by the change in deuterium labelled alanine in skin protein
Muscle mass | Baseline, 10 days
  Measured using Magnetic resonance imaging (MRI)
Body fat composition | Baseline, 10 days
  Measured using MRI
Resting energy expenditure | Baseline, 10 days
  Measured using indirect calorimetry
Systolic and diastolic blood pressure | Baseline, 5 days, 10 days
  Measured using automated device
Resting heart rate | Baseline, 5 days, 10 days
  Measured using automated device
Plasma amino acids | Baseline, 5 days, 10 days
  Measured in plasma samples
Blood metabolites | Baseline, 5 days, 10 days
  Assessed in plasma and serum samples
Urine metabolites | Baseline, 5 days, 10 days
  Measured in fasted urine samples
Skeletal muscle mitochondrial respiration | Baseline, 10 days
  Measured in skeletal muscle tissue collected from muscle biopsy
Skeletal muscle signalling pathways | Baseline, 10 days
  Measured in skeletal muscle tissue from muscle biopsy
Body mass | Baseline, 5 days, 10 days
  Assessed using scale
Dietary protein intake | 10 days
  Assessed by calculating the actual intakes from the provided diet
Dietary fat intake | 10 days
  Assessed by calculating the actual intakes from the provided diet
Dietary carbohydrate intake | 10 days
  Assessed by calculating the actual intakes from the provided diet
Liver fat | Baseline, 10 days
  Measured using MRI
Body lean mass composition | Baseline, 10 days
  Measured using MRI

OTHER OUTCOMES:
Age | Baseline
  At baseline, assessed using questionnaire
Height | Baseline
  Assessed using stadiometer

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands